CLINICAL TRIAL: NCT05516550
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Treamid in the Treatment of Patients With Persistent Lung Damage and Reduced Exercise Tolerance Following Acute Coronavirus Infection
Brief Title: Study to Assess Efficacy and Safety of Treamid for Patients With Reduced Exercise Tolerance After COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID-TRE-04
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV-2 Infection; Lung Fibrosis
Keywords: COVID-19; Tolerance to physical activity
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis | interventions — N,N'-bis(2-(1H-imidazol-2-yl)ethyl)pentanediamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A blind will be performed by using Placebo equivalent to Treamid tablets without active substance and the corresponding labeling of the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treamid 25 mg (Experimental): 1 tablet of Treamid 25 mg + 1 tablet of Placebo in the morning and 2 tablets of Placebo in the evening daily during 4 weeks of treatment period.
  Interventions: Drug: Treamid
- Treamid 50 mg twice a day (Experimental): 1 tablet of Treamid 25 mg + 1 tablet of Placebo in the morning and 1 tablet of Treamid 25 mg + 1 tablet of Placebo in the evening daily during 4 weeks of treatment period.
  Interventions: Drug: Treamid twice a day
- Treamid 50 mg once a day (Experimental): 2 tablets of Treamid 25 mg in the morning and 2 tablets of Placebo in the evening daily during 4 weeks of treatment period.
  Interventions: Drug: Treamid once a day
- Placebo (Placebo Comparator): 2 tablets of Placebo in the morning and 2 tablets of Placebo in the evening daily during 4 weeks of treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treamid — Participants will receive Treamid 25 mg once a day daily during 4 weeks
  Arms: Treamid 25 mg
Drug: Treamid twice a day — Participants will receive Treamid 25 mg in the morning and in the evening daily during 4 weeks
  Arms: Treamid 50 mg twice a day
Drug: Treamid once a day — Participants will receive Treamid 50 mg in the morning daily during 4 weeks
  Arms: Treamid 50 mg once a day
Drug: Placebo — Participants will receive Placebo in the morning and in the evening daily during 4 weeks
  Arms: Placebo

SUMMARY:
The innovative drug Treamid is planned for use in the treatment of patients with persistent lung damage and reduced exercise tolerance exertion after COVID-19 pneumonia in a multicenter, randomized, double-blind, placebo-controlled Phase IIb/III clinical study to assess the efficacy and safety of Treamid during a 28-day treatment.

The primary objective of the study is to prove that in the Treamid group, the proportion of patients achieving clinically significant load tolerance is statistically significantly higher than in the placebo group.

The secondary objective of the study is to evaluate the safety of Treamid and achievement of clinically significant improvements in indicators for various questionnaires and spirometry data.

DETAILED DESCRIPTION:
14-18 Russian centers are planned for participation in this study. The study consists of three periods: screening (2 weeks), treatment period (4 weeks) and follow-up period (4 weeks after completion of treatment with Treamid / Placebo).

412 patients with persistent lung damage and reduced exercise tolerance exertion after COVID-19 pneumonia are planned to be randomized.

Patients will be evaluated using the Modified British Medical Research Council (mMRC), six-minute walk test (6-MWT), Borg scale for dyspnea and fatigue, Dyspnea scale Index (BDI and TDI), KBILD questionnaire, EQ-5D-3L questionnaire, Hospital Anxiety and Depression Scale (HADS), Modified Fatigue Impact Scale (MFIS), Clinical Global Impression rating scales (CGI-I and CGI-S), chest computed tomography (CT), spirometry and body plethysmography with determination of DLCO.

All eligible patients will be randomized into 4 groups of 103 patients each in a 1:1:1:1 ratio: Treamid 25 mg in the morning and Placebo in the evening daily, Treamid 25 mg in the morning and Treamid 25 mg in the evening daily, Treamid 50 mg in the morning and Placebo in the evening daily, Placebo in the morning and Placebo in the evening daily. Patients will visit the study center at the Week 1, Week 2, Week 4 of treatment period and at the end of the follow up period. During all visits will be evaluated Adverse events (AEs), concomitant therapy, investigational drug registration, body weight, vital signs and Oxygen saturation (SpO2) scores. 6-MWT, Borg scale for dyspnea and fatigue, Dyspnea scale Index (TDI), KBILD questionnaire and MFIS will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Signed patient explanation sheet and informed consent for participation in the study.
2. Men and women at the age from 18 through 75 years old.
3. History of acute coronavirus infection:

   * The patient has a history of confirmed diagnosis of COVID-19 pneumonia, which resolved more than 2 weeks before screening;
   * History of COVID-19 is confirmed by positive qualitative analysis of SARS-CoV-2 by polymerase chain reaction (PCR) or detection of SARS-CoV-2 antigens;
   * Negative rapid test for SARS-CoV-2 antigen at screening and randomization;
   * Onset of first symptoms of COVID-19 from 42 to 120 days prior to randomization.
4. Severity of mMRC dyspnea ≥2 at screening and randomization.
5. Severity of exercise tolerance impairment at screening and randomization based on the 6-minute Walk Test:

   * reduction of the distance traveled below the normal limit (< 80% of predicted) at the level of shortness of breath ≥2 units according to the Borg scale;
   * severity of shortness of breath > 2 units according to the Borg scale, regardless of the presence of violations in the distance traveled.
6. The presence of foci of lung tissue seals such as "frosted glass" and/or interlobular septum seals, and/or areas of reticular changes in lung tissue, and/or the presence of areas (linear, focal) of lung tissue seals characteristic of COVID-19 confirmed by chest CT at screening. The percentage of lung tissue damage is ≥10%, but < 75% of the total lung volume.
7. The pulmonary diffusivity parameter is less than 80%, but more than 40% of predicted at the time of screening.
8. The patient's consent to use adequate contraception methods during the entire study and within 3 weeks after its completion. The adequate contraception methods include the use of the following:

   * oral or transdermal contraceptives;
   * condom or diaphragm (barrier method) with spermicide;
   * intrauterine device.

Exclusion Criteria:

1. Hypersensitivity to Treamid (active pharmaceutical substance XC268BG) and/or other components of the study drug.
2. History of invasive mechanical ventilation and high-flow oxygenation in the last 45 days or need for oxygen support at screening and randomization.
3. Chronic respiratory diseases diagnosed before COVID-19, including idiopathic pulmonary fibrosis and other interstitial lung diseases, moderate to severe bronchial asthma, moderate to severe chronic obstructive pulmonary disease, tuberculosis (including suspected tuberculosis based on CT examination at screening) or pulmonary hypertension.
4. Severe anemia (Haemoglobin < 70 g/L at screening).
5. Inability to perform a CT procedure (for example, a gypsum bandage or metal structures in the study area).
6. Severe cardiovascular disease at present or within 6 months prior to screening, including: Class III or IV chronic heart failure (New York Heart Association classification), clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation), unstable angina, myocardial infarction, heart and coronary vessel surgery, significant heart valve disease, uncontrolled hypertension with systolic blood pressure > 180 mmHg and diastolic blood pressure > 110 mmHg, pulmonary embolism arteries or deep vein thrombosis.
7. Chronic kidney disease or other significant kidney disease with glomerular filtration rate (GFR) < 60 mL/min (Cockcroft-Gault formula) at screening. Hemodialysis requirement at patient screening.
8. Stage II chronic liver failure (decompensated) and above; History of liver cirrhosis; alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) elevations of 3 or more times the upper limit of normal (ULN) at screening; increase in total bilirubin 2 or more times from ULN at screening (exception - Gilbert's syndrome in the history).
9. Severe diseases of the central nervous system, including a history of seizures or conditions that may lead to their development; stroke or transient ischemic attack within 6 months prior to screening; traumatic brain injury or loss of consciousness within 6 months prior to screening; brain tumor.
10. Malignancies requiring chemotherapy treatment within 5 years prior to screening or currently suspected cancer.
11. Participation in other clinical trials within 1.5 months prior to screening.
12. Requirement for or administration of the following drugs for 1 month prior to screening: erythropoietin, cytostatics, colchicine, cyclosporin A, interferon- γ -1b, bosentan, macitentan, etanercept, sildenafil, imatinib, warfarin, ambrisentan, nintedanib, pirfenidone, hyaluronidase asoxime 1 month prior to screening; glucocorticosteroids and N-acetylcysteine (requirement or 7 days prior to screening)
13. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption.
14. Signs of a marked uncontrolled concomitant disease, such as disorders of the nervous system, kidney, liver, endocrine system and gastrointestinal tract, which, in the opinion of the Investigator, could prevent the patient from participating in the study.
15. Positive test for human immunodeficiency virus (HIV), hepatitis B and/or C.
16. Alcohol or drug addiction, history of mental illness.
17. Severe, decompensated or unstable somatic diseases (any diseases or conditions that threaten the patient's life or impair the patient's prognosis, and make it impossible for him to participate in a clinical trial).
18. Patient's unwillingness or inability to comply with Protocol procedures (in the opinion of the study physician).
19. Pregnancy or breastfeeding period.
20. Other conditions that, in the opinion of the study physician, prevent the patient from entering the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically significant recovery of exercise tolerance (based on the 6MWD) from baseline values compared to Placebo. | Day 1- Day 29
  Clinically significant recovery of exercise tolerance is considered for patients with no significant abnormalities (Distance ≥ lower limit of normal), clinically significant decrease in the Borg dyspnea score (≥1 points), in the absence of a decrease in the distance traveled from the baseline values; for patients with severe abnormalities (Distance < lower limit of normal distance), clinically significant increase in the distance traveled by 54 or more meters with a decrease in the Borg dyspnea score (≥ 0.5 points) from the baseline values.

SECONDARY OUTCOMES:
Frequency of clinically significant change in lung diffusion capacity adjusted for hemoglobin (% of predicted) from baseline values compared to Placebo. | Day 1- Day 29
Rate of clinically significant recovery of exercise tolerance improvement using the Borg scale score at Visit 3, Visit 4, and Visit 5 from baseline values compared to Placebo. | Day 1- Day 56
Rate of clinically significant reduction in dyspnea by BDI/TDI scales at Visit 4 and Visit 5 from baseline values compared to Placebo. | Day 1- Day 56
Rate of clinically significant fatigue reduction assessed by change in MFIS fatigue score at Visit 4 and Visit 5 from baseline values compared to Placebo. | Day 1- Day 56
Rate of clinically significant reductions in Anxiety and Depression score assessed by HADS at Visit 4 and Visit 5 from baseline values compared to Placebo. | Day 1- Day 56
Rate of clinically significant increase in total KBILD score at Visit 4 and Visit 5 from baseline values compared to Placebo. | Day 1- Day 56
Rate of Clinically Significant Change in Patient Status on the Overall Clinical Impression Scale (CGI-S/CGI-I) at Visit 4 and Visit 5 from baseline values compared to Placebo. | Day 1- Day 56

OTHER OUTCOMES:
Rate of clinically significant recovery of exercise tolerance (based on the 6MWD) in female patients from baseline values compared to Placebo. | Day 1- Day 29
Change in DLCO according to bodyplethysmography at Week 4 relative to baseline values. | Day 1- Day 29
Change in Total Lung Capacity (TLC) according to bodyplethysmography at Week 4 relative to baseline. | Day 1- Day 29
The rate of reduction in the lung damage degree based on the computed tomography (CT) at Week 4 relative to the baseline value. | Day 1- Day 29
Mean Change in Lung Lesion (Expressed as % of Total Lung Area) by CT at Week 4 relative to the baseline value. | Day 1- Day 29
The rate of clinically significant increase in distance (54 or more meters) traveled within 6 minutes at Visit 3, Visit 4 and Visit 5 relative to the baseline value. | Day 1- Day 56
Mean change in distance traveled over 6 minutes at Visit 3, Visit 4 and Visit 5 (based on the 6MWD) relative to the baseline value. | Day 1- Day 56
Rate of clinically significant reduction in post-exercise dyspnea using the Borg scale score at Visit 3, Visit 4 and Visit 5 (based on the 6MWD) relative to the baseline value. | Day 1- Day 56
Mean change in post-exercise dyspnea using the Borg scale score at Visit 3, Visit 4 and Visit 5 (based on the 6MWD) relative to the baseline value. | Day 1- Day 56
Mean change in post-exercise fatigue using the Borg scale score at Visit 3, Visit 4 and Visit 5 (based on the 6MWD) relative to the baseline value. | Day 1- Day 56
Mean change in mMRC dyspnea severity at Visit 4 and Visit 5 relative to the baseline value. | Day 1- Day 56
Mean change in Anxiety and Depression score assessed by HADS at Visit 4 and Visit 5 relative to the baseline value. | Day 1- Day 56
Mean change from baseline in standardized health-related quality of life score assessed on the EQ-5D-3L scale at Visit 4 and Visit 5 relative to the baseline value. | Day 1- Day 56
Mean Change from Baseline in Total KBILD Score at Visit 3, Visit 4, and Visit 5 relative to the baseline value. | Day 1- Day 56
The rate of adverse events (AEs) | Day 1- Day 70
The rate of serious adverse events (SAEs) | Day 1- Day 70
Total number and proportion of patients with one or more AEs | Day 1- Day 70
Total number and proportion of patients who discontinued treatment due to AEs | Day 1- Day 70